CLINICAL TRIAL: NCT00447317
Title: Dietary Adherence Enhancement in Peritoneal Dialysis
Brief Title: Dietary Adherence Enhancement in Peritoneal Dialysis: BalanceWise-PD
Acronym: BalanceWise-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Mary Ann Sevick, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R21DK067181 (NIH)
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: End-Stage Renal Disease
Keywords: peritoneal dialysis; diet; sodium
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Intervention
  Interventions: Behavioral: BalanceWise-PD
- B (Other): Attention control, standard dietary education
  Interventions: Behavioral: Attention control

INTERVENTIONS:
Behavioral: BalanceWise-PD — Dietary counseling based on Social Cognitive Theory, paired with PDA-based dietary self-monitoring
  Arms: A
Behavioral: Attention control — Standard peritoneal dialysis dietary education
  Arms: B

SUMMARY:
This randomized study will pilot test an intervention, based on self-efficacy theory and involving personal digital assistant (PDA)-based dietary self-monitoring, to improve adherence to the peritoneal dialysis dietary regimen. 60 individuals, 21 years of age or older, who are on continuous ambulatory peritoneal dialysis or nightly cycler peritoneal dialysis, will be recruited to the study. Participants will be randomized to one of 2 groups. Group A will receive a 4-month active intervention of decreasing intensity over time delivered via mail, telephone, and during regularly scheduled dialysis clinic visits. Group B will receive a 4-month attention control experience in which they receive reinforcement of standard dietary education. With this study the investigators will:

1. Explore the impact of the intervention on dietary sodium intake,
2. Explore the intervention on blood pressure,
3. Explore the impact of the intervention on morning post dialysis weight (i.e. weight after conclusion of continuous cycling peritoneal dialysis (CCPD) or after long dwell for continuous ambulatory peritoneal dialysis (CAPD) patients, AND
4. Explore the feasibility and acceptability of the intervention

ELIGIBILITY:
Inclusion Criteria:

The investigators will recruit those individuals:

* who are 18 years of age or older,
* who are literate, community-dwelling adults, and
* who have been receiving maintenance PD for at least 3 months. Individuals on maintenance PD less than 3 months are excluded to allow for patients to adjust to the PD regimen, and for stabilization of nutritional status in the early weeks of dialysis (i.e. they may be considered for the study after 3 months of dialysis)

Exclusion Criteria:

Excluded from the study will be individuals:

* who are deemed by dialysis center staff to have a problem with cognitive function and to be chronically noncompliant to the dialysis regimen (e.g. misses multiple appointments and dialysis treatments),
* those who cannot read or write, those who do not speak English,
* those who plan to move out of the area or change dialysis centers within the next 5 months,
* those with a terminal illness and life expectancy of less than 12 months,
* those who are scheduled for a living donor transplant,
* individuals who cannot see the PDA screen or use the stylus to make selections from the PDA screen, or
* individuals who are living in a nursing home or personal care facility, who would have limited control over their dietary intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Dietary sodium intake as assessed from 3-day recalls. | baseline and 4 months
Dietary sodium effluent and urine concentration. | baseline and 4 months
Morning blood pressure. | baseline and 4 months
Morning post dialysis weight. | baseline and 4 months
Feasibility and acceptability of PDA-based dietary monitoring. | 4 months

SECONDARY OUTCOMES:
Dietary intake of protein, calories, and phosphorus. | baseline and 4 months
Perceived dietary barriers. | baseline and 4 months
Perceived dietary therapeutic efficacy. | baseline and 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Mary A Sevick, ScD, Principal Investigator — University of Pittsburgh
Locations (1):
- Dialysis Clinics, Inc., Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] McMahon EJ, Campbell KL, Bauer JD, Mudge DW, Kelly JT. Altered dietary salt intake for people with chronic kidney disease. Cochrane Database Syst Rev. 2021 Jun 24;6(6):CD010070. doi: 10.1002/14651858.CD010070.pub3. PMID 34164803